CLINICAL TRIAL: NCT01170013
Title: Substance Abuse Prevention for Preadolescents With Psychiatric Disorders
Brief Title: Substance Use Prevention in Teen Psychiatric Patients
Acronym: tCheckup
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21DA024207 (NIH)
Record Dates: First submitted 2010-06-02; First posted 2010-07-27 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Adolescent Substance Use
Keywords: substance use; adolescents; initiation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Check-up (Experimental): Two session motivational intervention to improve parent monitoring and communication with respect to adolescent risk behavior especially substance use
  Interventions: Behavioral: Family Check-up
- Psychoeducation (Active Comparator): Two sessions of psychoeducation for parents regarding adolescent risk behaviors especially substance use
  Interventions: Behavioral: Parent psychoeducation

INTERVENTIONS:
Behavioral: Family Check-up — Two session motivational intervention to improve parent monitoring and communication with respect to adolescent risk behavior especially substance use
  Other Names: Parent Motivational Interviewing
  Arms: Family Check-up
Behavioral: Parent psychoeducation — Two sessions of psychoeducation for parents regarding adolescent risk behaviors. especially substance use
  Other Names: Family psychoeducation
  Arms: Psychoeducation

SUMMARY:
The earlier a child initiates alcohol and other drug (AOD) use, the greater the risk of long-range problems. This association persists despite changes in national substance use rates over time, indicating its stability and viability as a target for prevention. At the same time, parent monitoring of youth behavior tends to decrease during the adolescent years, creating a source of risk for not only the early onset of AOD use but also escalation. Thus, programs are needed in parenting behaviors and family relationships that are protective in helping pre-adolescent youth to avoid initiation of AOD use and abuse. This is particularly true of children with psychiatric disorders who are at higher risk for developing AOD disorders than nonpsychiatrically disturbed children. The primary goal of this study is to test the effectiveness of a family-centered intervention to reduce the risk of AOD use among pre-adolescent children with a history of emotional/behavioral problems. In this application, the families of 80 youths aged 12-14 years, who have not yet begun AOD use but have been referred for mental health care due to psychiatric symptomatology, will be randomly assigned to receive either an individually tailored family program or standard care. The experimental intervention, which is based on the Family Check-Up model (Dishion & Kavanagh, 2003), provides a thorough assessment of family strengths and weaknesses as they relate to future risk for AOD use as well as emotional/behavioral problems, and utilizes principles of motivational interviewing to encourage families to change. Follow-up interviews will be conducted at 6 and 12 months after baseline to assess changes in parenting, AOD use, and other risky behaviors.

DETAILED DESCRIPTION:
The earlier a child initiates alcohol and other drug (AOD) use, the greater the risk of long-range problems. This association persists despite changes in national substance use rates over time, indicating its stability and viability as a target for prevention. At the same time, parent monitoring of youth behavior tends to decrease during the adolescent years, creating a source of risk for not only the early onset of AOD use but also escalation. Thus, programs are needed in parenting behaviors and family relationships that are protective in helping pre-adolescent youth to avoid initiation of AOD use and abuse. This is particularly true of children with psychiatric disorders who are at higher risk for developing AOD disorders than nonpsychiatrically disturbed children. The primary goal of this study is to test the effectiveness of a family-centered intervention to reduce the risk of AOD use among pre-adolescent children with a history of emotional/behavioral problems. In this application, the families of 80 youths aged 12-14 years, who have not yet begun AOD use but have been referred for mental health care due to psychiatric symptomatology, will be randomly assigned to receive either an individually tailored family program or standard care. The experimental intervention, which is based on the Family Check-Up model (Dishion & Kavanagh, 2003), provides a thorough assessment of family strengths and weaknesses as they relate to future risk for AOD use as well as emotional/behavioral problems, and utilizes principles of motivational interviewing to encourage families to change. Follow-up interviews will be conducted at 6 and 12 months after baseline to assess changes in parenting, AOD use, and other risky behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. the target child is between the ages of 12-14 years old at the start of the project and living at home with at least one parent/guardian
2. the target child must be receiving services at a mental health clinic and must screen in with a t- score of 70 or above on one of the DSM-oriented scales (ADHD, ODD, CD, anxiety problems, and affective problems) on the Child Behavior Checklist (i.e. reach the clinical cut-off)
3. the child must not report prior AOD use, and
4. parental consent and child assent are obtained.

Exclusion Criteria:

1. the target child is actively psychotic, and
2. the family is not able to speak and understand English or Spanish well enough to complete study procedures.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Parental monitoring/communication | 3 months
  Self-report and observational ratings of parent-child interactions with respect to limit setting, communication, and monitoring
Parental monitoring/communication | 6 months
  Self-report and observational ratings of parent-child interactions with respect to limit setting, communication, and monitoring

SECONDARY OUTCOMES:
marijuana use | 3 months
  frequency and quantity of marijuana use in the prior 30 days
marijuana use | 6 months
  frequency and quantity of marijuana use in the prior 30 days
alcohol use | 3 months
  frequency and quantity of alcohol use in the prior 30 days
alcohol use | 6 months
  frequency and quantity of alcohol use in the prior 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States